CLINICAL TRIAL: NCT04284982
Title: Periodized Resistance Training for Persistent Non-specific Low Back Pain: A Mixed Methods Feasibility Study
Brief Title: Periodized Resistance Training for Persistent Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/905
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Low Back Pain
Keywords: Exercise therapy; Resistance training
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heavy resistance training program (Experimental)
  Interventions: Behavioral: 16-week supervised heavy resistance training program with weekly undulating periodization

INTERVENTIONS:
Behavioral: 16-week supervised heavy resistance training program with weekly undulating periodization — Participants trained a whole-body program consisting of squat, bench press, deadlift and pendlay row two times per week for 16 weeks

SUMMARY:
In this study the feasibility is investigated of a 16-week supervised heavy resistance training program with weekly undulating periodization for individuals with persistent non-specific low-back pain.

ELIGIBILITY:
Inclusion Criteria:

* persistent non-specific low back pain with a duration >3 months
* average low back pain intensity last two weeks >= 4 on numerical pain rating scale (0-10 scale)
* no experience with heavy resistance training.

Exclusion Criteria:

* previous surgery of the low back
* radiculopathy
* structural spinal changes and/or specific spinal conditions that limit function (spinal stenosis, ankylosing spondylitis, spondylolisthesis/spondylolysis, protrusion, structural scoliosis)
* autoimmune and systemic inflammatory diseases
* cardiovascular disease
* neurological diseases
* severe osteoporosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Low back pain intensity on 0-10 Numerical Pain Rating Scale | 8 weeks
  From questionnaire: current pain, pain the last two weeks and pain the last four weeks, scale from 0-10 were 0 equals no pain and 10 equals the worst pain imaginable
Low back pain intensity on 0-10 Numerical Pain Rating Scale | 16 weeks
  From questionnaire: current pain, pain the last two weeks and pain the last four weeks, scale from 0-10 were 0 equals no pain and 10 equals the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Helbostad, prof, Study Director — Dept Neuromedicine and Movement Science, Fac MH, NTNU
Locations (1):
- Dept of Neuromedicine and Movement Science, Faculty of Medicine and Health Sciences, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Collected data and research protocol are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Tjosvoll SO, Mork PJ, Iversen VM, Rise MB, Fimland MS. Periodized resistance training for persistent non-specific low back pain: a mixed methods feasibility study. BMC Sports Sci Med Rehabil. 2020 May 8;12:30. doi: 10.1186/s13102-020-00181-0. eCollection 2020. PMID 32411374